CLINICAL TRIAL: NCT01389622
Title: Effect of Self-administered Auricular Acupressure on Smoking Cessation-a Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMC01
Record Dates: First submitted 2011-06-29; First posted 2011-07-08 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-03

CONDITIONS: Smoking Cessation
Keywords: Acupuncture; smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: NADA points and digital pressure (Experimental): Arm 1: NADA points and digital pressure with urge.
  Interventions: Other: acupuncture
- Arm 2: random points + digital pressure with urge (Experimental): Arm 2 (20 participants): random points + digital pressure with urge
  Interventions: Other: acupuncture
- Arm 3 (20 participants): NO acupressure, only advice + support (No Intervention)

INTERVENTIONS:
Other: acupuncture — National Acupuncture Detoxification Association (NADA) points + digital pressure
  Arms: Arm 1: NADA points and digital pressure
Other: acupuncture — random points + digital pressure
  Arms: Arm 2: random points + digital pressure with urge

SUMMARY:
Auricular acupressure has been practiced in China and Germany to help people in smoking cessation programs. The purpose of this clinical trial is to test for the clinical effectiveness of self-administered auricular acupressure as a non-invasive method for smoking cessation.

DETAILED DESCRIPTION:
Auricular acupressure has been practiced in China and Germany to help people in smoking cessation programs with varying degrees of success in different settings. The purpose of this clinical trial is to test for the clinical effectiveness of self-administered auricular acupressure as a non-invasive method for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Participants are included in the study if they satisfy the following criteria:

  * Male or female.
  * Between 18 and 75 years of age inclusive.
  * Able to provide informed consent to study.
  * History of tobacco cigarette smoking for at least 6 months.
  * Confirmed intention of smoking cessation with no more than 2 previous failed attempts in the last 3 year.

Exclusion Criteria:

* Existing pharmacotherapy for smoking cessation.
* History of major psychiatric disorder or chronic pain syndromes.
* More than 2 failed attempts of smoking cessation in the previous 3 years.
* History of other substance abuse.
* History of atopy, or suspected/known allergy to plaster.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Spot 7-day cessation rate | Weekly during the intervention period (weeks 1-6)
  Efficacy of intervention for smoking cessation

SECONDARY OUTCOMES:
Continuous Cessation Rate (CAR) | Weekly during the intervention period (weeks 1-6) and week 13 and week 26
  Efficacy of intervention for smoking cessation
End-expiratory carbon monoxide levels (CO) | Weekly during the intervention period (weeks 1-6) and week 13 and week 26
  Efficacy of intervention for smoking cessation
Adverse effects in terms of self-reported discomfort levels from auricular acupressure | Weekly during the intervention period (weeks 1-6)
  Nature and incidence of adverse events due to intervention
Stress level according to the Stress Check List (SCL) | Weekly during the intervention period (weeks 1-6) and week 13 and week 26
  Nature and incidence of adverse events due to intervention
Nicotine withdrawal symptoms according to Minnesota Nicotine Withdrawal Scale (MNWS) | Weekly during the intervention period (weeks 1-6) and week 13 and week 26
  Nature and incidence of adverse events due to intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Leung, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's Family Health Team, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Leung L, Neufeld T, Marin S. Effect of self-administered auricular acupressure on smoking cessation--a pilot study. BMC Complement Altern Med. 2012 Feb 28;12:11. doi: 10.1186/1472-6882-12-11. PMID 22373002